CLINICAL TRIAL: NCT03696810
Title: Characterization of Retinal Vascular Disease in Eyes With Mild to Moderate NPDR in Diabetes Type 2, Using Novel Non-invasive Imaging Methods, in a Longitudinal, Prospective and Interventional Clinical Study With 2 Years of Duration (CORDIS)
Brief Title: Characterization of Retinal Vascular Disease in Eyes With Mild to Moderate NPDR in Diabetes Type 2
Acronym: CORDIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEC/194/18
Record Dates: First submitted 2018-09-28; First posted 2018-10-05 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: NPDR - Non Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- • Laboratory tests (Other): • Laboratory tests (HbA1C levels and lipids)
  Interventions: Diagnostic Test: Laboratory tests

INTERVENTIONS:
Diagnostic Test: Laboratory tests — • Laboratory tests (HbA1C levels and lipids)

SUMMARY:
Characterization of Retinal vascular disease in eyes with mild to moderate NPDR in Diabetes type 2, using novel non-invasive Imaging methods, in a longitudinal, prospective and interventional clinical Study with 2 years of duration (CORDIS).

DETAILED DESCRIPTION:
Diabetic Retinopathy (DR) is a frequent complication of Diabetes Mellitus (DM) and is the main cause of vision loss in the working population in western countries.

Several studies provided evidence that good diabetic control is important to prevent and delay disease progression, but while some patients develop sight-threatening DR (STDR) despite good control, others escape the development of vison loss with poor metabolic control.

The STDR is defined as DME and PDR. DME is defined as thickening of the macula and is mainly due to accumulation of fluid in the central macular area resulting mainly from fluid leakage due to the alterations of the BRB. Identifying the eyes/patients at risk to develop central involved macular edema (CIME) and consequent vision-loss, as well as to understand its causes is fundamental for its appropriate treatment and, finally, to avoid vision loss due to DME.

Several studies have shown different prevalence's of DR, ranging from 10.1% to 48.1%.

The prevalence of DM in Portugal has increased and, between patients aged 20 to 79 years, was 11.7% in 2009, reaching 13.3% in 2013.

Chronic diseases often begin with a symptom-free phase being biomarkers fundamental in the identification of high-risk individuals in a reliably and timely manner, so that they can either be treated before onset of the disease or as soon as possible.

Our group has identified 3 different phenotypes of progression based on the microaneurysm (MA) turnover rate (sum of MA formation and disappearance rates) and central retinal thickness (RT) measurements obtained using non-invasive repeatable procedures: digital color fundus photography (CFP) and optical coherence tomography (OCT). MA turnover can identify eyes at risk of progression to Clinically Significant Macular Edema (CSME), as shown by our research results and an independent group. RT obtained with OCT provides insight into morphological changes of the retina in DR and DME, allowing the detection of retinal edema.

The current study will address only two of the published phenotypes, B and C, which show more rapid progression to STDR.

For an improved characterization of the main microvascular alterations that occur in NPDR, the investigators will use novel noninvasive, direct, objective and quantitative OCT-based methodologies: Optical coherence tomography angiography (OCTA) and OCT-Leakage (OCT-L).

OCTA allows the construction of three-dimensional blood flow information, and therefore can serve as a method to evaluate ocular circulation. OCTA is non-invasive and has the potential to be superior to fluorescein angiography (FA) in the detection and follow-up of DR lesions and mean vessel density measured in the superficial retinal layer in OCTA revealed to be a good differentiator between healthy eyes and eyes with DR. Vessel density was also correlated with best corrected visual acuity (BCVA) and severity of DR, suggesting that capillary closure may provide relevant information regarding progression of DR in individual patients with DM and may be a potential indicator for vision loss.

OCT-Leakage (OCT-L) is a new non-invasive imaging technique that performs automated analysis of the retinal extracellular space using spectral-domain optical coherence tomography (SD-OCT). Abnormal fluid accumulation is an indicator of breakdown of the blood-retinal barrier (BRB), which is an early and frequent finding in DR. Our research group showed the importance of this new method and demonstrated the increased sensitivity of OCT-L to detect abnormal fluid in the retina when compared with FA. This can be particularly useful to better characterize and identify features associated to leaky phenotype B.

A major objective of this study is to investigate changes in OCTA and OCT-L that may be biomarkers in the diagnosis and progression of NPDR and its ability to distinguish different stages of the disease. The identification with OCT-L of the abnormal fluid and alteration of the blood-retinal barrier (BRB), its location and quantification, complementing conventional OCTA, providing, therefore, information on capillary closure, vascular morphology and their alterations over 2 years, are expected to contribute to our understanding of DR progression.

Validation of biomarkers of DR progression, such as MA turnover and RT are important steps. However, OCTA and OCT-L offer an opportunity of improved characterization of the different DR phenotypes.

This study intends to better characterize the main alterations of the different phenotypes of DR considered to be leaky (OCT-L) or ischemic (OCTA), and to identify patients at risk of progression to STDR, identified in this study as central-involved ME (CIME), objectively measured by OCT or development of PDR, using these recent non-invasive techniques: OCTA and OCT-L.

ELIGIBILITY:
* Informed consent.
* Diabetes Mellitus type 2 according to 1985 WHO criteria.
* Age between 35 and 85 years.

At least in one eye:

Mild or moderate DR, with NPDR levels 20, 35, 43 and 47 (based on the ETDRS criteria - 7 fields CFP);

* Absence of CIME or PDR;
* Presence of at least 1 MA in the central 6000 µm in diameter area - Field 2;
* No previous intravitreal injections;
* BCVA 75 letters (20 /32);
* Refraction with a spherical equivalent less than 5 Dp.

At 6 months (Visit 2), at least one of the following criteria should be met:

Phenotype B criteria:

- OCT RT above the following thresholds (DRCR.net criteria)(16,29)

For ETDRS levels 20, 35, 43 and 47 at least 1 of the following criteria should be met at month 6:

Central RT (within centre circle 1000 µm in diameter area) above abnormal gender-specific thickness assessed based on OCT (DRCR.net criteria). Defined, considering Cirrus SD-OCT, the following thresholds (2):

* Central RT between 260 and 290 µm for women (SCME) and between 275 and 305 µm for men (SCME)
* Central RT greater than 290 µm for women (CIME) and Central RT greater than 305 µm for men (CIME).

OR

Phenotype C criteria:

- MA Turnover ≥ 6, assessed by RetmarkerDR. OR Patients who do not meet the eligibility criteria in visit 2 for phenotype B or C but that were previously identified as phenotype B or C will also be considered as eligible by investigator decision.

Exclusion Criteria

* Cataract or other eye disease that may interfere with fundus examinations.
* Glaucoma.
* Any eye surgery within a period of 6-months before the screening visit date.
* Other retinal vascular disease.
* Previous laser or intravitreal injection treatment.
* Dilatation of the pupil < 5 mm.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Development of CIME or PDR | 24 months
  Characterization of retinal microvascular changes occurring in eyes with mild to moderate NPDR
Capillary closure in the superficial and deep retinal vascular layers | 24 months
  Capillary closure in the superficial and deep retinal vascular layers by vessel density calculation, quantified by OCTA software (Angioplex, Zeiss);
LOR ratios | 24 months
  LOR ratios obtained with OCT-L analysis in the full retina and layer by layer.

SECONDARY OUTCOMES:
Microaneurysms turnover | 24 months
  Microaneurysms turnover computed from CFP using the RetmarkerDR software
Retinal Thickness | 24 months
  RT obtained with structural OCT in the full retina and by retinal layers

CONTACTS AND LOCATIONS:
Locations (1):
- AIBILI- Association for Biomedical Research and Inovation on Light and Image., Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marques IP, Ribeiro ML, Santos T, Reste-Ferreira D, Mendes L, Martinho AC, Santos AR, Figueira J, Lobo C, Cunha-Vaz J. Patterns of Progression of Nonproliferative Diabetic Retinopathy Using Non-Invasive Imaging. Transl Vis Sci Technol. 2024 May 1;13(5):22. doi: 10.1167/tvst.13.5.22. PMID 38780953